CLINICAL TRIAL: NCT02890914
Title: Transvaginal Ultrasound Training for the Obstetrics and Gynecology Resident: A Multi-Site Randomized Controlled Trial of Educational DVD
Brief Title: Transvaginal Ultrasound Training for Obstetrics and Gynecology Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: The Reading Hospital and Medical Center (Other); Main Line Health (Other)
Responsible Party: Principal Investigator, Rebekah McCurdy, MD, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 14E.231
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Ovarian Cysts
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Education (No Intervention): These residents received their standard residency education and experience.
- DVD Intervention (Experimental): These residents received a one-hour long DVD lecture in addition to standard residency education and experience.
  Interventions: Other: Transvaginal Ultrasound Educational DVD

INTERVENTIONS:
Other: Transvaginal Ultrasound Educational DVD — American Institute of Ultrasound in Medicine, "Gynecology: Beginners Only"®
  Arms: DVD Intervention

SUMMARY:
Obstetrics and gynecology residents are deemed to be proficient in transvaginal ultrasound (TVUS) upon graduation from an accredited program, although TVUS education in residency is not standardized. The objective of this study is to assess for improvement in transvaginal ultrasound knowledge among residents after viewing an educational DVD.

DETAILED DESCRIPTION:
This is a multi-site prospective parallel randomized controlled trial using an educational DVD from the American Institute of Ultrasound in Medicine, "Gynecology: Beginners Only"®, compared to routine education. All participants completed a pretest on transvaginal ultrasound images and principles. The intervention group repeated the test after viewing the DVD. During the trial, performing and logging transvaginal ultrasounds were encouraged. All enrolled residents repeated the test at 6-10 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* resident in obstetrics and gynecology at one of three sites

Exclusion Criteria:

* unable to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Difference in Pre and Post Study Mean Test Scores | 6-10 months

SECONDARY OUTCOMES:
Difference in Pre and Post Viewing Mean Test Scores | 1 hour
Difference in Number of Post-Study Logged Transvaginal Ultrasounds | Through study completion, an average of 2 years
Mean test score differences in specific question types (images and principles) | 6-10 months
Difference in mean scores on "orange cards" | 6-10 months

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah McCurdy, MD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein SR. Accreditation, certification: why all the confusion? Obstet Gynecol. 2007 Dec;110(6):1396-8. doi: 10.1097/01.AOG.0000289225.54215.e9. PMID 18055738
- [Background] Chao C, Chalouhi GE, Bouhanna P, Ville Y, Dommergues M. Randomized Clinical Trial of Virtual Reality Simulation Training for Transvaginal Gynecologic Ultrasound Skills. J Ultrasound Med. 2015 Sep;34(9):1663-7. doi: 10.7863/ultra.15.14.09063. Epub 2015 Aug 17. PMID 26283753
- [Background] Tolsgaard MG, Ringsted C, Dreisler E, Norgaard LN, Petersen JH, Madsen ME, Freiesleben NL, Sorensen JL, Tabor A. Sustained effect of simulation-based ultrasound training on clinical performance: a randomized trial. Ultrasound Obstet Gynecol. 2015 Sep;46(3):312-8. doi: 10.1002/uog.14780. Epub 2015 Aug 6. PMID 25580809
- [Background] Carolan-Rees G, Ray AF. The ScanTrainer obstetrics and gynaecology ultrasound virtual reality training simulator: A cost model to determine the cost viability of replacing clinical training with simulation training. Ultrasound. 2015 May;23(2):110-5. doi: 10.1177/1742271X14567498. Epub 2015 Jan 10. PMID 27433245